CLINICAL TRIAL: NCT01860768
Title: Potential Biomarkers for Early Diagnosis of Acute Aortic Dissection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, CHAI Xiangping, vice director of emergency department; vice director of hospital office, Central South University
Other Study IDs: 2XY-ED-001
Record Dates: First submitted 2013-05-04; First posted 2013-05-23 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Aortic Dissection; Biomarkers and Early Diagnosis
Keywords: Acute aortic dissection; Serum biomarkers; Early diagnosis
MeSH Terms: conditions — Aortic Dissection; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- acute aortic dissectin patients: definite diagnosis by computed tomography arteriography (CTA).
- acute chest pain patients: aortic dissection is exclude by aorta CTA

SUMMARY:
Acute aortic dissection (AAD) is an acute vascular lesions with high early misdiagnosis rate(31.8%), and mortality rate was 38%. In recent years, the incidence is rising and serious threat to human health. At present, the clinical diagnosis of AAD commonly used imaging methods, including chest X-ray, B ultrasound, CT, MRI and aortic angiography. Chest X-ray and two-dimensional ultrasound is limited in diagnosis of AAD, esophageal ultrasonography can display the intimal, identify the true and false lumen, but greater risk. CT, MRI and aortic angiography can be used as diagnosis method, but time-consuming, expensive and requires handling patients in emergency situations, should not be used as the preferred. Therefore, it is significance that biomarkers with high specificity and sensitivity for clinical fast diagnosis of AAD.

Parts small sample tests found that single serum α-smooth muscle actin (α-SMA), myosin heavy chain(MHC) and human soluble elastin fragments (sELAF) levels in patients with AAD were significantly higher than that of others (normal people, acute myocardial infarction patients). But because of the small study sample, limited control risk factors and incomplete comparison, their conclusions were questionable. In our previous studies also found that serum α-SMA, MHC and sELAF levels and the pathogenesis of AAD and prognosis are closely related. Therefore, on the basis, a prospective study is needed. We observe all the three biomarkers in enrolled patients with acute chest pain in emergency department, levels in healthy volunteers as the blank control. Then make definite diagnosis of the enrolled patients, and further observe the biomarkers dynamic change in AAD. Lastly, evaluate the early diagnostic value of combination serum α-SMA, MHC and sELAF level on patients with AAD.

DETAILED DESCRIPTION:
This is a prospective clinical study designed to procure blood samples from patients who present to the Emergency Department with suspected AAD.

Subjects enrolled in this study will sign and informed consent and have 3 blood samples drawn at different time points during their emergency department visit. In addition, data will be collected about the patient's health history, hospital procedures, and final diagnosis.

Blood samples collected in this study will be sent to laboratory for long-term storage and analysis in the future for these blood markers as they become available. No genetic testing will be conducted on these samples.

ELIGIBILITY:
Inclusion Criteria:

* chest pain without diagnosis confirmed
* symptom occurred in 2 hours
* ≥18 years old
* Can complete the base information
* Able and willing to give written consent

Exclusion Criteria:

* known AAD
* known causes of acute chest pain such as tumour and trauma
* pregnant or lactating female
* Associated chronic inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Alll patients presenting to the Second Xiangya Hospital of Central South Unversity Emergency Department with acute chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-02 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy(sensitivity and specificity of 400 participates for diagnosing acute aortic dissection) of serum biomarkers on patients with AAD. | 1 day (Emergency room without follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China